Analysis plan: PRODICA, Maria Hedelin Version 2

# Statistical analysis plan

Identifiers: NCT02759380

Brief Title: Can Dietary Phytoestrogens Slow Down Prostate Tumor Proliferation? (PRODICA)

Official Title: Can Dietary Phytoestrogens Slow Down Prostate Tumor Proliferation? A

Randomized Study (PRODICA)

Principal Investigator: Maria Hedelin

Date: 2022-05-31

#### AIM

The overall aim of the PRODICA-study is to increase the knowledge, for the impact of diet on prostate tumor proliferation.

#### **HYPOTHESIS**

- In men diagnosed with intermediate risk-level prostate cancer, the addition of phytoestrogenrich foods containing 200 mg phytoestrogens per day in six weeks, gives a reduced prostate tumor proliferation compared to an absence of the addition of phytoestrogen-rich foods during the same period.
- 2) If the effect of phytoestrogens on prostate tumor proliferation exists, it is modified by a SNP in the promoter region of the estrogen-beta-gene (rs 2987983-13950).

## STUDY DESIGN

The study design is shown in Figure 1. Men diagnosed with intermediate-risk prostate cancer T1–T2 (Gleason score <8, PSA <20), scheduled for radical prostatectomy, are identified at the Sahlgrenska University Hospital. Interested men are contacted by phone and a first meeting is scheduled. At the meeting the participants receive verbal and written information and sign an informed consent. A food frequency questionnaire including dietary and living habits and supplements are filled in and baseline blood samples are taken. The men are randomized to a diet or a control group through a closed envelop. All participants receive general dietary advice according to the Swedish National Food Agency (1). Participants are instructed to avoid supplements but no other dietary restrictions are given. The diet group receive a food package including food items high in phytoestrogens. Recipes and serving suggestions for the study diet are also given. The intake of the food items gradually steps up according to a schedule and the items are eaten in specific amounts until the surgery.

The participants are contacted by phone once during the study and a 24-hour recall is performed. The interview is made to control compliance in the study group and to estimate the intake of phytoestrogens in the control group. Near to surgery a similar food frequency questionnaire is filled in and endpoint blood samples are taken. Prostate biopsies are taken at the surgery. Hormones and PSA are analyzed from baseline and endpoint blood samples. The expression of androgen receptor and estrogen receptor alfa and beta are analyzed in tumor material. Tumor proliferation is calculated by ki-67 from prostatectomy specimens at surgery.



## NUMBER OF SUBJECTS

The person time studied will be 203 person moments. Interim analyzes will be made when there is data to analyze 100 person moments.

#### **INCLUSION CRITERIA**

- Patients with prostate cancer T1–T2, Gleason score <8, prostate-specific antigen (PSA) <20
- scheduled for radical prostatectomy.

## **EXCLUSION CRITERIA**

Ongoing hormone therapy
Difficult physical or psychological conditions or diminished cognitive function
Allergy or intolerance of the intervention foods

#### **DATA MANAGEMENT**

## **Definition of primary outcome**

#### Ki-67

Tumor proliferation rate (Ki-67) is measured in prostatectomy specimens from the surgery. The ratio of stained prostate cancer nuclei is calculated in five different areas and the median, mean, and max

values are calculated

Analyze of prostatectomy specimens from the surgery, variables:

ki67\_median (median value of ki-67)

**ki67** mean (mean value of ki-67)

**ki67** max (max value of ki-67)

Above variables will be dichotomized according to the median value in the study

population:ki67\_median\_cat (0/1)

ki67 mean cat (0/1)

ki67 max cat (0/1)

## **Definition of secondary outcomes**

Levels of PSA are analyzed from blood samples taken at the inclusion meeting (baseline) and in connection with another visit within one week before surgery (endpoint). The difference is calculated between endpoint and baseline.

#### **PSA**

**PSA\_total\_BL** (total PSA levels at baseline)

**PSA total EP** (total PSA levels at endpoint)

**PSA total diff** (difference in total PSA levels, endpoint-baseline)

**PSA total diff cat** (total PSA difference endpoint-baseline, decreased/unchanged=0, increased=1)

**PSA** ratio BL (PSA ratio free/total at baseline)

PSA ratio EP (PSA ratio free/total at endpoint)

PSA ratio diff (difference in total PSA levels, endpoint-baseline)

PSA ratio diff cat (PSA ratio diff endpoint-baseline, decreased/unchanged=0, increased=1))

#### Hormones

Concentrations of testosterone, estradiol, sex hormone binding globulin

(SHBG), and IGF-1 will be analyzed in serum at endpoint and baseline. The difference is calculated between endpoint and baseline.

**Estradiol BL** (Estradiol levels at baseline)

Estradiol\_EP (Estradiol levels at endpoint)

Estradiol diff (difference in Estradiol levels, endpoint-baseline)

estradiol diff cat (Estradiol difference endpoint-baseline, decreased/unchanged=0, increased=1)

**Testosterone BL** (Testosterone levels at baseline)

**Testosterone** EP (Testosterone levels at endpoint)

**Testosteron\_diff** (difference in Testosteron levels, endpoint-baseline)

testo diff cat (Testosteron difference endpoint-baseline, decreased/unchanged=0, increased=1)

IGF1\_BL (IGF1 levels at baseline)

**IGF1 EP** (IGF1 levels at endpoint)

**IGF1** difference (difference in IGF1 levels, endpoint-baseline)

**SHBG BL** (SHBG levels at baseline)

**SHBG** EP (SHBG levels at endpoint)

**SHBG\_difference** (difference in SHBG levels, endpoint-baseline)

**testo\_estrad\_ratio\_diff** (ratio testosterone/estradiol difference endpoint-baseline) **testo\_SHBG\_ratio\_diff** (ratio testosterone/SHBG difference endpoint-baseline)

## Gene expression

The radical prostatectomy tissues are collected at surgery and formalin fixed paraffin embedded. Expression of genes involved in proliferation and ER signal pathways and cell-cycle progression (CCP) gene expression will be analyzed to identify the expression of genes involved in tumorigenesis. Global transcriptome-wide expression array Clariom D® will be used. For analysis of the CCP score, gene expression of the genes involved in CCP based on the Prolaris® gene panel and the Decipher Score. Thereafter, guided and unguided analyses will be performed.

## Receptors expression

One benign- and one cancer biopsies are collected at surgery.  $ER\alpha$ ,  $ER\beta$ , and AR mRNA expression will be determined.

**ER\_a** (mRNA levels of estrogen receptor  $\alpha$ )

**ER\_b** (mRNA levels of estrogen receptor  $\beta$ )

**AR** (mRNA levels of androgen receptor)

#### **Definition of exposure**

The participants in the intervention group are defined as exposed and the participants in the control group are defined as not exposed.

**Group intervention** (0=control, 1=intervention)

Intake of different phytoestrogens at endpoint is based on information from the Food Frequency Questionnaire (FFQ) and the 24-h dietary recall.

**Phytoestogens\_EP\_3** (intake of phytoestrogens at endpoint divided in tertiles, calculated from the FFO)

**Lignans EP 3** (intake of lignans at endpoint divided in tertiles, calculated from the FFQ)

**Isoflavones** EP 3 (intake of isoflavones at endpoint divided in tertiles, calculated from the FFQ)

Coumestrol N58 EP 2 (dichotomized intake of coumesterol at endpoint, calculated from the FFQ)

Phyto 24 recall 3 (intake of phytoestrogens at the 24-h dietary recall divided in tertiles)

The concentrations of phytoestrogens (daidzein, enterodiol, enterolactone, equol, genistein, glycetein,

lariciresinol, and secoisolariciresinol) in plasma for a sub-group of participants:

**lignans\_EP\_nmol** (plasma levels of lignans at endpoint=enterolactone+ enterodiol+ lariciresinol+ seco EP nmol)

**lignans\_BL\_nmol** ((plasma levels of lignans at baseline=enterolactone+ enterodiol+ lariciresinol+ seco EP nmol)

**isoflavones\_EP\_nmol** (plasma levels of isoflavones at endpoint = daidzein\_EP\_nmol + genistein EP nmol + glycitein EP nmol + equol EP nmol)

**isoflavones\_BL\_nmol** (plasma levels of isoflavones at baseline = daidzein\_EP\_nmol + genistein EP nmol + glycitein EP nmol + equol EP nmol)

phytoestrogens\_EP\_nmol (plasma levels of total phytoestrogens at baseline =
enterolactone\_EP\_nmol + enterodiol\_EP\_nmol + lariciresinol\_EP\_nmol + seco\_EP\_nmol +
daidzein\_EP\_nmol + genistein\_EP\_nmol + glycitein\_EP\_nmol + equol\_EP\_nmol)

phytoestrogens\_BL\_nmol (plasma levels of total phytoestrogens at endpoint =
enterolactone\_BL\_nmol + enterodiol\_BL\_nmol + lariciresinol\_BL\_nmol + seco\_BL\_nmol +
daidzein BL nmol + genistein BL nmol + glycitein BL nmol + equol BL nmol)

lignans diff nmol = lignans EP nmol - lignans BL nmol

isoflav\_diff\_nmol= isoflavones\_EP\_nmol - isoflavones\_BL\_nmol

phyto diff nmol= phytoestrogens EP nmol - phytoestrogens BL nmol

## Definition of effect modifying factor

The individual genotype (alleles TT, TC or CC) of the estrogen-beta-gene (ERB) are identified in the blood sample at baseline.

cat genotype (created from variable Genotype, 0=TT, 1= TT/CC)

#### PLANS FOR STATISTICAL ANALYZES

## VARIABLES TO ANALYZE

Created variables (for more details see attached variable list):

```
BMI (kg/m²):
BMI_stata = Weight_inclusion / ((Lenght_inclusion/100) * (Lenght_inclusion/100)
BMI_group = 1= under weight (BMI <18.5); 2= normal weight (BMI 18.5-24.9); 3= Overweight (BMI 25-29.9); 4= Obese class (BMI 30-34.9) 1; 5= Obese class ≥2 (BMI ≥35)
Weight change (kg):
Weight diff = Weight endpoint - Weight inclusion
```

Compliance (1= compliance  $\ge$ 80; 0= compliance <80 %):

Compliance 24 recall (based on reported intake of phytoestrogens at the 24-h dietary recall)

Compliance\_intervention\_24\_r (based on eaten interventions foods reported from at the 24-h dietary recall)

Compliance\_intervention (based on eaten interventions foods reported from at the end of the intervention)

Intake of isoflavones (µg):

Isoflavones\_ BL = Genistein\_N56\_BL + Daidzein\_N57\_BL + Formononetin\_N59\_BL + Biochanin N60 BL + Equol N75 BL

Isoflavones\_EP = GenisteinN56\_EP + Daidzein\_N57\_EP + Formononetin\_N59\_EP + Biochanin N60 EP + Equal N75 EP.

Intake of lignans (µg):

Lignans\_BL = SECOtot\_N61\_BL + Matairesinol\_N62\_BL Lariciresinol\_N71\_BL + Pinoresinol\_N72\_BL + Syringaresinol\_N73\_BL + Medioresinol\_N74\_BL + Enterodiol\_N76\_BL + Enterolactone N77\_BL

Lignans\_EP=SECOtot\_N61\_EP + Matairesinol\_N62\_EP + Lariciresinol\_N71\_EP + Pinoresinol\_N72\_EP + Syringaresinol\_N73\_EP + Medioresinol\_N74\_EP + Enterodiol\_N76\_EP + Enterolactone N77\_EP

Intake of phytoestrogens (ug):

Phytoestogens\_BL = (Isoflavones\_BL + Lignans\_BL + Coumestrol\_N58\_BL) Phytoestogens EP =(Isoflavones EP + Lignans EP + Coumestrol\_N58\_EP)

Level of physical activity:

Physical activity BL group = low, moderate or high

1 = Low physical activity (101, 102, 103 or 201 points)

2 = Moderate physical activity (104, 202, 203, 301 or 302 points)

3 = High physical activity (204, 303, 304, 401, 402, 403 or 404 points)

Intake of fatty fish:

Fat\_fish\_group\_BL: 0 = <1 times/month; 1 = 1-3 times/month;  $2 = \ge 1$  times/week Fat\_fish\_group\_EP: 0 = <1 times/month; 1 = 1-3 times/month;  $2 = \ge 1$  times/week Fat fish diff: Fat fish month EP - Fat fish month BL

Use of antibiotics:

antiobotics\_1y\_dic (0= no intake last year or don't know;  $1=\ge 1$  time last year) antiobotics\_2\_5y\_dic (0= no intake last 2-5 years or don't know;  $1=\ge 1$  time last 2-5 years) f53\_1\_EP: Intake of antibiotics in recent weeks at endpoint (0= No; 1=Yes) antibiotics\_all (0= no intake during intervention and last 5 years or don't know;  $1=\ge 1$  time during intervention and last 5 years)

Smoking:

0= never smoked or quitted smoking >5 years ago

1= Current smoker or quitted smoking ≤5 years ago

#### STATISTICAL MODELS

Difference between groups will be tested for variables stated below. Independent T-test or Mann-Whitney U-test will be used for continuous variables depending on if the data has a normal or skewed distribution. Fishers's exact test will be used for categorical variables.

## Covariates to test (possible confounding factors):

- Energy\_kcal\_EP\_3 (total energy intake at endpoint, categorized in tertiles)
- Sum\_satured\_fat\_EP\_3 (sum of saturated fats (g) at endpoint, categorized in tertiles)
- Fat fish group EP (categorized intake of fat fish at endpoint)
- Calcium EP 3 (intake of calcium at endpoint, categorized in tertiles)
- Physical activity BL group (categorized physical activity at baseline)
- f47 1 EP (changed physical activity during intervention)
- Biopsies\_cancer (percent of biopsies with cancer at diagnosis)
- gleason cat (categorized Gleason score at diagnosis)
- gleason cat rp (categorized Gleason score at surgery)
- rp teritargradjanej (categorized tertiary Gleason degree at surgery)
- Age inclusion (continuous age at baseline)
- BMI group (BMI at baseline in groups)
- Weight diff (difference in weight between endpoint and baseline)
- smoking (categorized smoking at baseline)
- heredity (categorized heredity at baseline)
- Zinc EP 3 (intake of zinc at endpoint, categorized in tertiles)
- Alcohol EP 3 (intake of alcohol at endpoint, categorized in tertiles)
- Sum\_monosat\_fat\_EP\_3 (intake of monounsaturated fatty acids at endpoint, categorized in tertiles)
- Sum\_polysat\_fat\_EP\_3 (intake of polyunsaturated fatty acids at endpoint, categorized in tertiles)
- red meat EP 3 (intake of red meat at endpoint, categorized in tertiles)
- vegetables all EP 3 (intake of vegetables at endpoint, categorized in tertiles)
- fruit\_all\_EP\_3 (intake of fruits at endpoint, categorized in tertiles)
- Vit\_E\_EP\_3 (intake of vitamin E at endpoint, categorized in tertiles)

• Finasteride (intake of Finasteride under intervention, no=0, yes=1)

Pearson or Spearman correlation coefficient will be used to evaluate whether dietary covariates are correlated. If the correlation coefficient between two covariates in the model or between covariates and the main exposure are higher than 0.6, multicolinearity issues is considered, eventually one of the covariates will be excluded from the model.

## Model building:

The association between intake of phytoestrogens and tumor proliferation will evaluated by regression models, providing estimate of risk difference (RD) relative risk (RR) and corresponding 95% confidence intervals.

#### Crude models:

## C0: Ki-67

C1: C0 + Group intervention

C2: C0 + Phytoestogens\_EP

C3: C0 + Isoflavones EP

C4: C0 + Lignans EP

C5: C0 + Coumestrol N58 EP

## C0<sub>2</sub>: PSA total diff

C1<sub>2</sub>: C0<sub>2</sub> + Group intervention

C2<sub>2</sub>: C0<sub>2</sub> + Phytoestogens EP

C3<sub>2</sub>: C0<sub>2</sub> + Isoflavones EP

C4<sub>2</sub>: C0<sub>2</sub> + Lignans EP

C5<sub>2</sub>: C0<sub>2</sub> + Coumestrol N58 EP

## C03: PSA ratio diff

 $C1_3$ :  $C0_3$  + Group intervention

C3<sub>3</sub>: C0<sub>3</sub> + Phytoestogens EP

C4<sub>3</sub>: C0<sub>3</sub> + Isoflavones EP

C5<sub>3</sub>: C0<sub>3</sub> + Lignans EP

C6<sub>3</sub>: C0<sub>3</sub> + Coumestrol N58 EP

### C0<sub>4</sub>: estradiol diff cat

C14: C04 + Group\_intervention

C3<sub>4</sub>: C0<sub>4</sub> + Phytoestogens EP

## Analysis plan: PRODICA, Maria Hedelin

Version 2

C4<sub>4</sub>: C0<sub>4</sub> + Isoflavones EP

C5<sub>4</sub>: C0<sub>4</sub> + Lignans EP

C6<sub>4</sub>: C0<sub>4</sub> + Coumestrol N58 EP

C05: testo diff cat

C1<sub>5</sub>: C0<sub>5</sub> + Group intervention

C3<sub>5</sub>: C0<sub>5</sub> + Phytoestogens EP

C4<sub>5</sub>: C0<sub>5</sub> + Isoflavones EP

C5<sub>5</sub>: C0<sub>5</sub> + Lignans EP

C6<sub>5</sub>: C0<sub>5</sub> + Coumestrol N58 EP

C06: testo estrad ratio diff

C1<sub>6</sub>: C0<sub>6</sub> + Group intervention

C3<sub>6</sub>: C0<sub>6</sub> + Phytoestogens EP

C4<sub>6</sub>: C0<sub>6</sub> + Isoflavones EP

C5<sub>6</sub>: C0<sub>6</sub> + Lignans EP

C6<sub>6</sub>: C0<sub>6</sub> + Coumestrol N58 EP

C07: testo SHBG ratio diff

C<sub>17</sub>: C<sub>07</sub> + Group intervention

C3<sub>7</sub>: C0<sub>7</sub> + Phytoestogens EP

C4<sub>7</sub>: C0<sub>7</sub> + Isoflavones EP

C57: C07 + Lignans EP

 $C6_7$ :  $C0_7$  + Coumestrol\_N58\_EP

## Final model:

Which covariates included in the model will be based on:

- 1) If a known risk factor for the outcome (based on previous subject matter knowledge and with the help of Directed Acyclic Graphs)
- 2) If differs between groups of exposure
- 3) proportional ( $\geq 10\%$ ) change in  $\beta$ -coefficients

## Stratification by ERB alleles and test of interaction:

Analysis of hypothesis above (C0- C07 and corresponding models) will be stratified by genotype of

ERβ (variable: cat genotype).

Interactions between exposure and ERB SNPs on the outcome will be evaluated on the additive effect scales. Effects will be measured by RDs and interaction will be assessed in a generalized linear model by the product term between the covariates representing phytoestrogen intake and SNP genotypes.

Product term: int1=intervention\*cat genotype

## **Additional analysis:**

*Intention-to-treat-analyses*: All participants will be included.

*Per-protocol-analyzes*: All participants with ≥80 % compliance will be included.

In the intervention group, compliance will be considered as  $\ge 80$  percent of the recommended intake of 200 mg of phytoestrogens, which is equal to  $\ge 160$  mg. In the control group, intakes below 160 mg of phytoestrogens will be considered compliant.

Analysis of hypothesis will be stratified for:

- no use of antibiotics vs. use of antibiotics
- no use of finasteride vs. use of finasteride

Investigate the effects of the intervention diet on plasma concentrations of phytoestrogens: Cohen's Kappa will be used to compare the agreement of classifications in tertiles from estimated intake of phytoestrogens and plasma concentrations of phytoestrogens. (Kappa values <0 will be considered as poor, 0.00-0.20 as slight, 0.21-0.40 as fair, 0.41-0.60 as moderate, 0.61-0.80 as substantial, and 0.81-1.00 as almost perfect). Boxplots will be used to present the data graphically. Linear regressions will be used to investigate the relationships between estimated intake concentrations (explanatory variables) and plasma concentrations of phytoestrogens (outcomes). The regression model will be stratified according to the intervention- and control groups and genotype.

## Receptor expression

The mRNA levels of ER $\alpha$ , ER $\beta$ , and AR will be compared between intervention- and control groups and groups of genotype.

## **AUTHORS**

Rebecca Ahlin, rebecca.ahlin@vgregion.se, 076-618 5020

Maria Hedelin, maria.hedelin@oncology.gu.se, 070-7401858

#### REFERENCES

1. Livsmedelsverket. Kostråden - hitta ditt sätt. [2018-03-07 cited]; Available from: <a href="https://www.livsmedelsverket.se/matvanor-halsa--miljo/kostrad-och-matvanor/rad-om-bra-mat-hitta-ditt-satt/">https://www.livsmedelsverket.se/matvanor-halsa--miljo/kostrad-och-matvanor/rad-om-bra-mat-hitta-ditt-satt/</a>.

| Analysis plan: PRODICA, Maria Hedelin | Version 2 |
|---------------------------------------|-----------|

## **APPENDICES**

Appendics 1 - Variable list

Appendics 2 - Food Frequency Questionnaire